CLINICAL TRIAL: NCT04211844
Title: Metabolic Changes in Chronic Hepatitis C Virus Patients Receiving Direct Acting Antivirals
Brief Title: Metabolic Changes in Chronic HCV Patients Receiving DAAS
Acronym: HCV DAAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nehal Khaled Abdel Raouf Abdel Fattah, Principal Investigator, Ain Shams University
Other Study IDs: 164
Record Dates: First submitted 2019-11-26; First posted 2019-12-26 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Sofosbuvir; daclatasvir; ledipasvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sofosbuvir plus daclatasvir: 50 patients receiving 400 mg sofosbuvir plus daclatasvir 60 mg once daily for 12 weeks. Blood samples are taken at baseline (week 0), week 4 (during treatment) and week 24 (post treatment after discontinuation of treatment at sustained virological response). Samples will be evaluated for lipid profiles, fasting blood sugar and glycated hemoglobin.
  Interventions: Drug: sofosbuvir plus daclatasvir
- sofosbuvir plus ledipasvir: 50 patients receiving 400 mg sofosbuvir plus ledipasvir 90 mg (Harvoni) once daily for 12 weeks. Blood samples are taken at baseline (week 0), week 4 (during treatment) and week 24 (post treatment after discontinuation of treatment at sustained virological response). Samples will be evaluated for lipid profiles, fasting blood sugar and glycated hemoglobin.
  Interventions: Drug: Sofosbuvir plus Ledipasvir

INTERVENTIONS:
Drug: sofosbuvir plus daclatasvir — 50 patients in the first group will receive 400 mg sofosbuvir plus daclatasvir 60 mg once daily for 12 weeks.
  Other Names: Sovaldi Daklinza
  Groups: sofosbuvir plus daclatasvir
Drug: Sofosbuvir plus Ledipasvir — 50 patients in the second group will receive 400 mg sofosbuvir plus ledipasvir 90 mg (Harvoni) once daily for 12 weeks.
  Other Names: Harvoni
  Groups: sofosbuvir plus ledipasvir

SUMMARY:
Observational Study to check metabolic changes between two different hepatitis C antiviral medication groups. This study will evaluate the impact of different treatments on Serum lipid changes, fasting blood glucose and glycated hemoglobin . It will determine if changes are due to different Antiviral regimens or due to different Sustained virological response rates.

DETAILED DESCRIPTION:
The aim of this study is;

* To investigate and compare the changes in the total lipid profile and glycated hemoglobin (HbA1c) for chronic hepatitis C patients after receiving either one of two different direct antiviral regimens: sofosbuvir/daclatasvir and sofosbuvir/ledipasvir (Harvoni).
* To evaluate the impact of treatment response on the serial changes of serum lipid levels and glycated hemoglobin after receiving either of the two different direct antiviral regimens.
* To determine whether the change in the lipid profile and HbA1C is due to different antiviral regimens or due to different SVR rates.

Recruitment will be based on reviewing newly admitted patients and choosing those who are treatment naive and easy to treat according to study inclusion criteria. Thorough check of patient file will be done before starting the study. Eligible patients will sign a consent before starting both the treatment and the study. Patients will be divided into two groups taking treatment for 12 weeks. After treatment, patients will be followed-up for up to 12 weeks.

Patients will be asked to fast for a total of 12 hours. First 8 hours of fasting, a blood sample will be withdrawn for fasting blood sugar and glycated hemoglobin. At 12 hours of fasting, another sample will be withdrawn for lipid profile.

At baseline, patients dermographics (sex, age, weight, height, BMI), full medication history and full medical history will be collected from both patient file and patient consultation. After end of treatment at week 24, weight will be measured and BMI will be also be calculated. Adverse effects reporting:Patients will be asked about any undesirable effects detected throughout the trial which would be reported.

For the whole study period, patients will be subjected to assessment of the following:

* CBC, ALT, AST, total serum bilirubin, and creatinine will be done every 4 weeks (week 0, 4, 8, 12, 16, and 24)
* Complete lipid profile, fasting blood glucose, and HbA1c levels at baseline, during therapy (week 4), and at week 24 after discontinuation of therapy.
* Quantitative PCR for HCV RNA at week 0 and 24.

Results will be collected and tabulated in excel sheet to undergo statistical analysis. Statistical analyses will be done using the SPSS software (Statistical Package for the Social Sciences). Proportions will be compared using Fisher's exact test and means will be compared with Student's t-test or Wilcoxon rank sum test, where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 18 to 75 years old. Patients ≥ 65 years old should undergo cardiological assessment prior to therapy by ECG, echocardiography and cardiological consultaion.
* Easy to treat group: treatment naïve patients with serum HCV RNA positivity by PCR.
* Clinically stable condition.
* Platelet count ≥ 150,000/mm³.
* INR ≤ 1.2
* Serum albumin ≥ 3.5 g/dl.
* Total serum bilirubin ≤ 1.2 mg/dl.
* eGFR > 30 ml/min

Exclusion Criteria:

* Pregnancy or inability to use effective contraceptives.
* Inadequately controlled diabetes mellitus (HbA1c > 9%)
* HCV-HIV co infection.
* HBV-HCV co infection.
* Any cause for chronic liver disease other than hepatitis C
* Hyper or hypothyroidism.
* Hepatocellular carcinoma, except 6 months after intervention aiming at cure with no evidence of activity by dynamic imaging (CT or MRI)
* Extra-hepatic malignancy except after two years of disease-free interval.
* Fibrosis: FIB-4 index ≥ 3
* Patients prescribed with lipid-lowering agents (statins).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cases involved in the study will be recruited from El-Demerdash Ain Shams University Hospital in Cairo, Egypt. Patients will be followed up at the "HCV treatment unit Ain Shams University Hospital" for the whole study period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Total Lipid Profile within 6 months | baseline, week 4 (during treatment), week 24 (after end of treatment)
  serum cholesterol, High density lipoproteins, Low density lipoproteins, Triglycerides, very low density lipoprotein , all measured in mg/dL after 12 hours of fasting
Change from baseline Glycosylated Hemoglobin within 6 months | baseline, week 4 (during treatment), week 24 (after end of treatment)
  average level of blood sugar over the past 2 to 3 months, measured in percentage %
Change from baseline Fasting Blood Glucose within 6 months | baseline, week 4 (during treatment), week 24 (after end of treatment)
  measured as mg/DL after 8 hours of fasting

SECONDARY OUTCOMES:
Treatment Response | 12 WEEKS after end of therapy
  Sustained Virological Response at week 12 after end of treatment ( SVR 12)

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Abdel Fattah, PharmB, Principal Investigator — Ain Shams University
Locations (1):
- El Demerdash Hospital, Cairo, Abbasseya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.